CLINICAL TRIAL: NCT00352378
Title: A Phase III Randomized Study of Primary Chemotherapy With Adriamycin/Cyclophosphamide(AC) vs Taxotere/Xeloda(TX) for Stage II and III Breast Cancer
Brief Title: Primary Chemotherapy With Adriamycin/Cyclophosphamide(AC) vs Taxotere/Xeloda(TX) for Stage II and III Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Jungsil Ro / Center for Breast Cancer, National Cancer Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-02-034
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2007-09

CONDITIONS: Breast Cancer
Keywords: Primary
MeSH Terms: conditions — Breast Neoplasms | interventions — Anthracyclines; Cyclophosphamide; Docetaxel; Capecitabine; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adriamycin plus Cyclophosphamide (Experimental): Intravenous infusion of Adriamycin 60mg/m2 , over 30 min, onD1 and Intravenous infusion of cyclophosphamide 600 mg/m2 over 30 min on D1.
  Interventions: Drug: Anthracycline, Cyclophosphamide, Docetaxel, Capecitabine
- Taxotere plus Xeloda (Experimental): Intravenous infusion of Taxotere 75 mg/m2 over 1 hr, on D1, and Xeloda 1000mg/m2.p.o. BID x 14days on D1-D14
  Interventions: Drug: Anthracycline, Cyclophosphamide, Docetaxel, Capecitabine

INTERVENTIONS:
Drug: Anthracycline, Cyclophosphamide, Docetaxel, Capecitabine — Patients will be randomized to receive regimen A (AC) and regimen B(TX),preoperatively as follows:
  Regimen A (AC): Intravenous infusion of Adriamycin 60mg/m2 , over 30 min, onD1 and Intravenous infusion of cyclophosphamide 600 mg/m2 over 30 min on D1. Regimen B(TX): Intravenous infusion of Taxotere 75 mg/m2 over 1 hr, on D1, and Xeloda 1000mg/m2.p.o. BID x 14days on D1-D14
  Other Names: Taxotere; Xeloda; Cytoxan; doxorubicin

SUMMARY:
This is an open labeled phase III randomized trial. The patients with clinical stage II and III will undergo mammotome biopsy of breast tumor for histologic diagnosis, immunohistochemical studies for estrogen receptor(ER), progesterone receptor(PR), HER-2/neu and others. PET results will determine the positivity of lymph node metastasis.

DETAILED DESCRIPTION:
- Patients will be randomized to receive regimen A (AC) and regimen B(TX), preoperatively,as follows: Regimen A (AC): Intravenous infusion of Adriamycin 60mg/m2 , over 30 min, onD1 and Intravenous infusion of cyclophosphamide 600 mg/m2 over 30 min on D1. Regimen B(TX): Intravenous infusion of Taxotere 75 mg/m2 over 1 hr, on D1, and Xeloda 1000mg/m2.p.o. BID x 14days on D1-D14 The cycle repeats every 3 weeks for 4 times. Premedication for regimen A includes antiemetics, for regimen B, dexamethasone as routinely given.

Patients who do not respond to the initial two cycles of preoperative chemotherapy will undergo operation.

The response rate will be determined by the number of patients with complete and partial responses according to RECIST guidelines. Pathologic complete response is defined as no pathologic evidence of residual disease. Safety will be evaluated by the frequency, severity, and relationship of adverse events graded by NCI Common Toxicity Criteria(CTC) that occur during the treatment and follow-up periods. Time to disease progression will be calculated from the date of study entry to the first objective documentation of progressive disease. Response duration will be measured from the date a patient first fulfills the CR or PR criteria to the first date of objective documentation of disease progression. Survival time will be calculated from the date of study entry to the date of death

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologically confirmed and newly diagnosed breast cancer: stage II and III breast cancer.
* PET results will determine node positivity.
* No prior hormonal , chemotherapy or radiotherapy is allowed.
* No breast operation other than biopsy to make diagnosis is allowed.
* Age:18-years and older, not pregnant pre-, and postmenopausal women with good performance status (ECOG 0-1)
* Adequate hematopoietic function:

  1. Absolute granulocyte count >=1500/mm3,
  2. platelet >=100,000/mm3, Hemoglobin >=10 g/mm3
* Adequate renal function: Serum creatinine <=1.5 mg/dl
* Adequate hepatic function:

  1. total bilirubin: <=1.5 mg/dl
  2. AST/ALT: <=three times normal
  3. Alkaline phosphatase: <=three times normal
* Adequate cardiac function: normal or nonspecific EKG taken within 1 mo of enrollment

Exclusion Criteria:

* Patients who received hormonal , chemotherapy or radiotherapy for breast cancer
* Patients who underwent surgery for breast cancer
* Patients who have history of cancer other than in situ uterine cervix cancer or nonmelanotic skin cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2002-06; Primary Completion 2005-10 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
pathologic complete remission | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jungsil Ro, MD,PhD, Principal Investigator — National Cancer Center, Korea